CLINICAL TRIAL: NCT02510560
Title: A Multi-center, Double-blind, Randomized, Three-Arm, Parallel-Group, Placebo Controlled Study to Assess the Efficacy and Safety of NTRA-2112 on Intestinal Malabsorption in Preterm Infants
Brief Title: Study to Assess the Efficacy and Safety of NTRA-2112 on Intestinal Malabsorption in Preterm Infants
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Elgan Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIT-04
Record Dates: First submitted 2015-07-24; First posted 2015-07-29 (Estimated); Results first posted 2025-06-06 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Premature Birth of Newborn; Intestinal Malabsorption
MeSH Terms: conditions — Premature Birth; Malabsorption Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NTRA-2112 A (Experimental): NTRA-2112 A - Dose 1 To be administered orally with daily feed for 28 days or until discharge from hospital.
  Interventions: Drug: NTRA-2112
- NTRA-2112 B (Experimental): NTRA-2112 B - Dose 2 To be administered orally with daily feed for 28 days or until discharge from hospital.
  Interventions: Drug: NTRA-2112
- Placebo (Placebo Comparator): Placebo To be administered orally with daily feed for 28 days or until discharge from hospital.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NTRA-2112
  Arms: NTRA-2112 A; NTRA-2112 B
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study will evaluate the effect of NTRA-2112 on intestinal malabsorption in preterm infants.

DETAILED DESCRIPTION:
The study will assess the efficacy and safety of NTRA-2112 on intestinal malabsorption in preterm infants as compared to placebo

ELIGIBILITY:
Inclusion Criteria

1. Male or female pre-term infant 26 and up to 32 weeks gestation. Gestational age matching (±2 weeks) between maternal dates and/or early antenatal ultrasound
2. Birth weight ≥ 500g
3. Singleton or twin birth

Exclusion Criteria

1. Complete enteral feeding

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2016-10-09 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (4):
  - Vidant Medical Center, Greenville, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Belgium (5):
  - AZ Sint-Jan, Bruges
  - UZ Brussel, Brussels
  - CHR de la Citadelle, Liège
  - CHC Cliniques Saint-Vincent, Rocourt
  - GZA Sint-Augustinus, Wilrijk
- France (3):
  - CHRU Nancy, Maternité Régionale, Nancy
  - CHU Necker-Enfants Malades, Paris
  - CHU - Hôpital Sud, Rennes
- Germany (5):
  - Kinderklinik, Evangelisches Waldkrankenhaus Spandau, Berlin
  - Klinik und Poliklinik fur Kinder-und Jugendmedizin, Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Klinik fur Neugeborene, Kinder und Jugendliche, Universitatsklinik der Paracelsus Medizinischen Privatuniversitat, Nuremberg
  - Klinik fuer Kinder und Jugendliche, Helios Klinikum Pforzheim, Pforzheim
  - Kinderklinik, Evangelisches Waldkrankenhaus, Spandau
- Hungary (4):
  - DE KK Gyermekklinika, Debrecen
  - Szegedi Tudomanyegyetem Szent Gyorgyi Albert Klinikai Kozpont Gyermekgyogyaszati klinika Koraszulott Intenzív Osztaly, Szeged
  - Fejéktató Kórhz Újszülött, Csecsemő és Gyermekosztály - Megyei Szent György Egyetemi, Székesfehérvár
  - Csolnoky Ferenc Korhaz, Veszprém
- Israel (8):
  - Barzilai MC, Ashkelon
  - Soroka Medical Center, Beersheba
  - Bnai Zion MC, Haifa
  - Rambam Health Care Campus, Haifa
  - Laniado, Netanya
  - Schneider Children's Medical Center, Petah Tikva
  - Sheba MC, Ramat Gan
  - Tel Aviv Sourasky MC, Tel Aviv
- Italy (7):
  - Presidio Ospedaliero G. Salesi - AOUI Ospedali Riuniti di Ancona, Ancona
  - Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale dei Bambini "V.Buzzi"- Azienda ICP, Milan
  - Azienda Ospedaliera San Gerardo, Monza
  - Policlinico Gemelli, Rome
  - Azienda Ospedaliero Universitaria, Udine
  - Ospedale F. Del Ponte - Azienda Ospedaliera di Varese, Varese
- Netherlands (3):
  - AMC - Academic Medical Center, Amsterdam
  - UMC Groningen (UMCG), Beatrix Kinderziekenhuis, Groningen
  - Isala Klinieken, Zwolle
- Spain (6):
  - Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - La-Paz, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - CHUS - Complejo Hospitalario Universitario de Santiago, Santiago
  - Hospital Universitario La Fe, Valencia
- United Kingdom (5):
  - Bradford Royal Infirmary, Bradford
  - University Hospital of Leicester NHS Trust- Royal Infirmary, Leicester
  - Queen's Medical College, Nottingham
  - Queens Medical Center, Nottingham
  - Portsmouth Hospitals NHS Trust, Portsmouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mank E, Saenz de Pipaon M, Lapillonne A, Carnielli VP, Senterre T, Shamir R, van Toledo L, van Goudoever JB; FIT-04 Study Group. Efficacy and Safety of Enteral Recombinant Human Insulin in Preterm Infants: A Randomized Clinical Trial. JAMA Pediatr. 2022 May 1;176(5):452-460. doi: 10.1001/jamapediatrics.2022.0020. PMID 35226099

RESULTS

PARTICIPANT FLOW:
Groups:
- NTRA-2112 A: NTRA-2112 A - Dose 1 To be administered orally with daily feed for 28 days or until discharge from hospital.
  NTRA-2112
- NTRA-2112 B: NTRA-2112 B - Dose 2 To be administered orally with daily feed for 28 days or until discharge from hospital.
  NTRA-2112
- Placebo: Placebo To be administered orally with daily feed for 28 days or until discharge from hospital.
  Placebo
Period: Overall Study
Arm/Group | NTRA-2112 A | NTRA-2112 B | Placebo
Started | 108 | 94 | 98
Completed | 77 | 72 | 76
Not Completed | 31 | 22 | 22
Not completed — Discontinued from Treatment | 27 | 18 | 19
Not completed — Other | 4 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Due to early study termination by the Sponsor, only 300 of the 450 intended subjects were enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | NTRA-2112 A | NTRA-2112 B | Placebo | Total
Number analyzed (Participants) | 108 | 94 | 98 | 300
Age, Customized [Count of Participants; unit: Participants]
  26-28 weeks | 49 | 46 | 51 | 146
  29-32 weeks | 58 | 48 | 47 | 153
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 51 | 54 | 169
  Male | 44 | 43 | 44 | 131
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 6 | 17
  White | 78 | 72 | 69 | 219
  More than one race | 24 | 17 | 22 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 25 | 24 | 25 | 74
  Belgium | 14 | 5 | 8 | 27
  Hungary | 7 | 6 | 5 | 18
  United States | 6 | 5 | 5 | 16
  Italy | 15 | 13 | 15 | 43
  United Kingdom | 5 | 3 | 5 | 13
  Israel | 9 | 6 | 8 | 23
  France | 4 | 10 | 12 | 26
  Germany | 3 | 2 | 2 | 7
  Spain | 17 | 19 | 11 | 47
  Bulgaria | 3 | 1 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Days to Achieve Complete Enteral Feeding
Description: Numbers of days to achieve full enteral feeding (NFE) is defined as:
  Number of Days to the first day of achieving enteral feeding of at least 150 ml/kg/day, which must be sustained for at least 3 consecutive days.
Time Frame: 28 days or discharge from hospital
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NTRA-2112 A | NTRA-2112 B | Placebo
Number analyzed (Participants) | 84 | 78 | 76
Days | 9.3 (4.81) | 10.0 (6.09) | 10.3 (5.10)
Statistical Analysis 1: Comparison: NTRA-2112 A vs Placebo; Test type: Superiority; p = 0.115, Stratified Van Elteren Test
Statistical Analysis 2: Comparison: NTRA-2112 B vs Placebo; Test type: Superiority; p = 0.243, Stratified Van Elteren Test

2. Secondary Outcome: Number of Days to Achieve Discharge From Hospital or Readiness to Discharge
Description: Readiness for discharge from hospital is defined as achieving all of the below:
  * Infant weight ≥ 1800g
  * Stable body temperature
  * Capable of oral feeding (reached full enteral feeding and not dependent on PN)
Time Frame: 28 days or discharge from hospital
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NTRA-2112 A | NTRA-2112 B | Placebo
Number analyzed (Participants) | 87 | 82 | 85
Days | 36.4 (16.26) | 33.8 (14.36) | 36 (15.21)
Statistical Analysis 1: Comparison: NTRA-2112 A vs Placebo; Test type: Superiority; p = 0.714, Stratified Van Elteren Test
Statistical Analysis 2: Comparison: NTRA-2112 B vs Placebo; Test type: Superiority; p = 0.243, Stratified Van Elteren Test

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | NTRA-2112 A | NTRA-2112 B | Placebo
All-Cause Mortality (participants affected / at risk) | 5/108 | 1/88 | 4/97
Serious Adverse Events (participants affected / at risk) | 15/108 | 10/88 | 19/97
Other Adverse Events (participants affected / at risk) | 91/108 | 70/88 | 81/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NTRA-2112 A (N=108) | NTRA-2112 B (N=88) | Placebo (N=97)
Anaemia neonatal (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 | 3 | 1
Cystic fibrosis (Congenital, familial and genetic disorders) | 1 | 0 | 0
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 7 | 3 | 8
Necrotising colitis (Gastrointestinal disorders) | 0 | 1 | 3
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Ileal stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Neonatal gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Injury associated with device (General disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Sepsis neonatal (Infections and infestations) | 4 | 2 | 5
Neonatal pneumonia (Infections and infestations) | 0 | 0 | 2
Meningitis neonatal (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Systemic candida (Infections and infestations) | 1 | 0 | 0
subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 | 1 | 0
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Neonatal respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
patent ductus arteriosus repair (Surgical and medical procedures) | 1 | 1 | 0
Hypertension neonatal (Vascular disorders) | 0 | 0 | 1
Iliac vein occulsion (Vascular disorders) | 1 | 0 | 0
Neonatal hypotension (Vascular disorders) | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NTRA-2112 A (N=108) | NTRA-2112 B (N=88) | Placebo (N=97)
Anaemia neonatal (Blood and lymphatic system disorders) | 39 | 34 | 34
Anaemia (Blood and lymphatic system disorders) | 18 | 14 | 13
Bradycardia neonatal (Cardiac disorders) | 6 | 2 | 3
Neonatal tachycardia (Cardiac disorders) | 3 | 5 | 1
patent ductus arteriosis (Congenital, familial and genetic disorders) | 12 | 9 | 9
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 7 | 3 | 8
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 5 | 5
Sepsis neonatal (Infections and infestations) | 9 | 6 | 8
Ophthalmia neonatorum (Infections and infestations) | 4 | 6 | 10
Neonatal hyponatraemia (Metabolism and nutrition disorders) | 12 | 8 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 5 | 3
Intraventricular haemorrhage neonatal (Nervous system disorders) | 3 | 5 | 2
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 4 | 4 | 5
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 12 | 16
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 2
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 3
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT02510560/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT02510560/SAP_001.pdf